CLINICAL TRIAL: NCT01290887
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Reslizumab (3.0 mg/kg) as Treatment for Patients With Eosinophilic Asthma Who Completed a Prior Teva-Sponsored Study in Eosinophilic Asthma
Brief Title: Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Reslizumab (3.0 mg/kg) as Treatment for Patients (12 Through 75 Years of Age) With Eosinophilic Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C38072/3085; 2010-024540-15 (EudraCT Number)
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — reslizumab; Antibodies, Monoclonal, Humanized

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reslizumab 3.0 mg/kg (Experimental): Reslizumab 3.0 mg/kg administered intravenously once every 4 weeks ( +-7 days) for up to 24 months.
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — Reslizumab (3.0 mg/kg) administered intravenously by infusion every 28 days (±7 days), for approximately 24 months
  Other Names: Cinquil; humanized monoclonal antibody; CEP-38072

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of reslizumab at a dosage of 3.0 mg/kg every 4 weeks for approximately 24 months in pediatric and adult patients with eosinophilic asthma as assessed by adverse events, physical examination findings, vital sign measurements, and concomitant medication usage throughout the study (every 4 weeks), clinical laboratory test results, and measurement of antidrug antibodies.

DETAILED DESCRIPTION:
Study patients deemed eligible based on activities from the preceding Teva sponsored double blind study of reslizumab in eosinophilic asthma. Specifically, as per inclusion criterion c, patients must have either completed treatment in a previous Teva-sponsored study or have received at least 2 doses of study drug treatment in a pulmonary function study.

Eligible patients could enroll in this study only after completion of the end of treatment visit in a Teva sponsored, randomized, placebo controlled, double blind study of reslizumab in eosinophilic asthma, which served as the screening/baseline visit for participation in this open label extension study. The use of systemic corticosteroids for asthma in any of the previous Teva sponsored double blind studies of reslizumab did not exclude patients from this study. The previous Teva studies were C38072/3081 (NCT01270464), C38072/3082 (NCT01287039), and C38072/3083 (NCT01285323).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* Patient must have completed treatment in a previous Cephalon-sponsored double-blind asthma exacerbation study or received at least 2 doses of study drug treatment in a pulmonary function study.
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.
* other criteria may apply; please contact the investigator for more information.

Exclusion Criteria:

* The patient has a clinically meaningful comorbidity that would interfere with the study schedule or procedures, or compromise the patient's safety.
* The patient has another confounding underlying lung disorder (eg, chronic obstructive pulmonary disease, pulmonary fibrosis, or lung cancer).
* The patient is a current smoker.
* The patient is expected to be poorly compliant with study drug administration, study procedures, or visits.
* The patient has any aggravating factors that are inadequately controlled (e.g., gastroesophageal reflux disease [GERD]).
* Female patients who are pregnant, or nursing, or, if of childbearing potential and not using a medically accepted, effective method of birth control (eg, spermicide, abstinence, intrauterine device [IUD], or steroidal contraceptive [oral, transdermal, implanted, and injected] in conjunction with a barrier method) are excluded from this study.
* The patient has a current infection or disease that may preclude assessment of asthma.
* other criteria may apply; please contact the investigator for more information.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Senior Director - Worldwide Clinical Research, Study Director — Cephalon
Locations (219):
- United States (48):
  - Teva Investigational Site 58, Scottsdale, Arizona
  - Teva Investigational Site 12, Anaheim, California
  - Teva Investigational Site 11, Fountain Valley, California
  - Teva Investigational Site 41, Fresno, California
  - Teva Investigational Site 59, Long Beach, California
  - Teva Investigational Site 43, Los Angeles, California
  - Teva Investigational Site 4, Orange, California
  - Teva Investigational Site 15, Walnut Creek, California
  - Teva Investigational Site 2, Colorado Springs, Colorado
  - Teva Investigational Site 34, Colorado Springs, Colorado
  - Teva Investigational Site 47, Denver, Colorado
  - Teva Investigational Site 28, Waterbury, Connecticut
  - Teva Investigational Site 53, Clearwater, Florida
  - Teva Investigational Site 24, Largo, Florida
  - Teva Investigational Site 27, Miami, Florida
  - Teva Investigational Site 55, Miami, Florida
  - Teva Investigational Site 5, Miami, Florida
  - Teva Investigational Site 52, Orlando, Florida
  - Teva Investigational Site 19, Tallahassee, Florida
  - Teva Investigational Site 17, Trinity, Florida
  - Teva Investigational Site 18, Valrico, Florida
  - Teva Investigational Site 25, Lawrenceville, Georgia
  - Teva Investigational Site 6, Lilburn, Georgia
  - Teva Investigational Site 3, Savannah, Georgia
  - Teva Investigational Site 49, Lexington, Kentucky
  - Teva Investigational Site 46, Bangor, Maine
  - Teva Investigational Site 40, St Louis, Missouri
  - Teva Investigational Site 74, St Louis, Missouri
  - Teva Investigational Site 64, Boys Town, Nebraska
  - Teva Investigational Site 8, Omaha, Nebraska
  - Teva Investigational Site 26, Summit, New Jersey
  - Teva Investigational Site 30, Winston-Salem, North Carolina
  - Teva Investigational Site 20, Cincinnati, Ohio
  - Teva Investigational Site 31, Cincinnati, Ohio
  - Teva Investigational Site 50, Oklahoma City, Oklahoma
  - Teva Investigational Site 1, Medford, Oregon
  - Teva Investigational Site 66, Altoona, Pennsylvania
  - Teva Investigational Site 73, Lincoln, Rhode Island
  - Teva Investigational Site 9, Providence, Rhode Island
  - Teva Investigational Site 21, Charleston, South Carolina
  - Teva Investigational Site 32, Nashville, Tennessee
  - Teva Investigational Site 63, Boerne, Texas
  - Teva Investigational Site 44, Dallas, Texas
  - Teva Investigational Site 69, El Paso, Texas
  - Teva Investigational Site 16, Fort Worth, Texas
  - Teva Investigational Site 14, San Antonio, Texas
  - Teva Investigational Site 45, San Antonio, Texas
  - Teva Investigational Site 33, Madison, Wisconsin
- Argentina (8):
  - Teva Investigational Site 121, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 126, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 127, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 128, Quilmes-Buenos Aires
  - Teva Investigational Site 125, Rosario
  - Teva Investigational Site 123, Rosario-Santa Fe
  - Teva Investigational Site 120, San Miguel de Tucuman - Tucuma
  - Teva Investigational Site 122, San Miguel de Tucuman - Tucuma
- Australia (4):
  - Teva Investigational Site 641, East Bentleigh
  - Teva Investigational Site 642, Frankston
  - Teva Investigational Site 645, Liverpool
  - Teva Investigational Site 643, Nedlands
- Belgium (5):
  - Teva Investigational Site 261, Brussels
  - Teva Investigational Site 264, Brussels
  - Teva Investigational Site 260, Ghent
  - Teva Investigational Site 262, Jambes
  - Teva Investigational Site 263, Liège
- Brazil (7):
  - Teva Investigational Site 146, Belo Horizonte
  - Teva Investigational Site 150, Florianópolis
  - Teva Investigational Site 140, Porto Alegre
  - Teva Investigational Site 144, Porto Alegre
  - Teva Investigational Site 147, Porto Alegre - RS
  - Teva Investigational Site 143, Porto Alegre, RS
  - Teva Investigational Site 142, Santo André
- Canada (4):
  - Teva Investigational Site 103, Calgary
  - Teva Investigational Site 101, Montreal
  - Teva Investigational Site 104, Newmarket
  - Teva Investigational Site 105, Windsor
- Chile (5):
  - Teva Investigational Site 160, Rancagua
  - Teva Investigational Site 164, Santiago
  - Teva Investigational Site 161, Temuco
  - Teva Investigational Site 162, Valdivia
  - Teva Investigational Site 166, Valparaíso
- Colombia (4):
  - Teva Investigational Site 181, Bogotá
  - Teva Investigational Site 185, Bogotá
  - Teva Investigational Site 182, Cali
  - Teva Investigational Site 180, Floridablanca
- Czechia (7):
  - Teva Investigational Site 287, Brno
  - Teva Investigational Site 284, Břeclav
  - Teva Investigational Site 286, Liberec
  - Teva Investigational Site 280, Olomouc
  - Teva Investigational Site 281, Olomouc
  - Teva Investigational Site 285, Olomouc
  - Teva Investigational Site 283, Tábor
- Teva Investigational Site 300, Odense, Denmark
- France (2):
  - Teva Investigational Site 342, Marseille
  - Teva Investigational Site 341, Montpellier
- Germany (8):
  - Teva Investigational Site 361, Berlin
  - Teva Investigational Site 366, Berlin
  - Teva Investigational Site 371, Bochum
  - Teva Investigational Site 369, Frankfurt
  - Teva Investigational Site 370, Hamburg
  - Teva Investigational Site 372, Koblenz
  - Teva Investigational Site 367, Leipzig
  - Teva Investigational Site 363, Mainz
- Teva Investigational Site 380, Athens, Greece
- Hungary (7):
  - Teva Investigational Site 401, Balassagyarmat
  - Teva Investigational Site 400, Miskolc
  - Teva Investigational Site 404, Mosonmagyaróvár
  - Teva Investigational Site 403, Sopron
  - Teva Investigational Site 407, Százhalombatta
  - Teva Investigational Site 402, Tatabánya
  - Teva Investigational Site 405, Törökbálint
- Israel (9):
  - Teva Investigational Site 423, Ashkelon
  - Teva Investigational Site 432, Haifa
  - Teva Investigational Site 425, Jerusalem
  - Teva Investigational Site 428, Jerusalem
  - Teva Investigational Site 426, Kfar Saba
  - Teva Investigational Site 422, Petah Tikva
  - Teva Investigational Site 433, Ramat Gan
  - Teva Investigational Site 421, Rehovot
  - Teva Investigational Site 420, Tel Aviv
- Malaysia (5):
  - Teva Investigational Site 705, Batu Caves
  - Teva Investigational Site 701, George Town
  - Teva Investigational Site 700, Kuala Lumpur
  - Teva Investigational Site 702, Kuala Lumpur
  - Teva Investigational Site 704, Taiping
- Mexico (7):
  - Teva Investigational Site 203, Distrito Federal
  - Teva Investigational Site 204, Guadalajara, JAL
  - Teva Investigational Site 200, Hermosillo, Sonora
  - Teva Investigational Site 205, Mexico City
  - Teva Investigational Site 207, Mexico City
  - Teva Investigational Site 209, Monterrey
  - Teva Investigational Site 202, Tijuana, B.C.
- Teva Investigational Site 460, Heerlen, Netherlands
- New Zealand (5):
  - Teva Investigational Site 723, Auckland
  - Teva Investigational Site 724, Dunedin
  - Teva Investigational Site 727, Hamilton
  - Teva Investigational Site 720, Tauranga
  - Teva Investigational Site 721, Wellington
- Peru (8):
  - Teva Investigational Site 223, Cercado de Lima, Lima
  - Teva Investigational Site 220, Lima
  - Teva Investigational Site 221, Lima
  - Teva Investigational Site 222, Lima
  - Teva Investigational Site 225, Lima
  - Teva Investigational Site 226, Lima
  - Teva Investigational Site 227, Lima
  - Teva Investigational Site 229, Lima
- Philippines (5):
  - Teva Investigational Site 742, Manila
  - Teva Investigational Site 740, Quezon City
  - Teva Investigational Site 741, Quezon City
  - Teva Investigational Site 743, Quezon City
  - Teva Investigational Site 745, Quezon City
- Poland (8):
  - Teva Investigational Site 507, Bialystok
  - Teva Investigational Site 509, Bydgoszcz
  - Teva Investigational Site 513, Gdansk
  - Teva Investigational Site 512, Lodz
  - Teva Investigational Site 505, Lublin
  - Teva Investigational Site 500, Ostrów Wielkopolski
  - Teva Investigational Site 511, Poznan
  - Teva Investigational Site 504, Tarnów
- Romania (5):
  - Teva Investigational Site 523, Bucharest
  - Teva Investigational Site 524, Bucharest
  - Teva Investigational Site 520, Cluj-Napoca
  - Teva Investigational Site 521, Iași
  - Teva Investigational Site 522, Târgu Mureş
- Russia (14):
  - Teva Investigational Site 545, Barnaul
  - Teva Investigational Site 549, Kemerovo
  - Teva Investigational Site 543, Moscow
  - Teva Investigational Site 544, Moscow
  - Teva Investigational Site 554, Moscow
  - Teva Investigational Site 558, Moscow
  - Teva Investigational Site 559, Moscow
  - Teva Investigational Site 555, Novosibirsk
  - Teva Investigational Site 557, Novosibirsk
  - Teva Investigational Site 540, Saint Petersburg
  - Teva Investigational Site 541, Saint Petersburg
  - Teva Investigational Site 542, Saint Petersburg
  - Teva Investigational Site 552, Tomsk
  - Teva Investigational Site 546, Yaroslavl
- Slovakia (4):
  - Teva Investigational Site 563, Bradejov
  - Teva Investigational Site 561, Levice
  - Teva Investigational Site 560, Spišská Nová Ves
  - Teva Investigational Site 562, Topoľčany
- South Africa (9):
  - Teva Investigational Site 584, Cape Town
  - Teva Investigational Site 586, Cape Town
  - Teva Investigational Site 587, Centurion
  - Teva Investigational Site 582, Durban
  - Teva Investigational Site 585, Durban
  - Teva Investigational Site 580, Johannesburg
  - Teva Investigational Site 589, Johannesburg
  - Teva Investigational Site 583, Pretoria
  - Teva Investigational Site 588, Pretoria
- South Korea (6):
  - Teva Investigational Site 682, Gwangju
  - Teva Investigational Site 680, Seoul
  - Teva Investigational Site 681, Seoul
  - Teva Investigational Site 683, Seoul
  - Teva Investigational Site 686, Seoul
  - Teva Investigational Site 685, Suwon
- Sweden (5):
  - Teva Investigational Site 602, Gothenburg
  - Teva Investigational Site 604, Gothenburg
  - Teva Investigational Site 603, Linköping
  - Teva Investigational Site 600, Lund
  - Teva Investigational Site 601, Malmo
- Taiwan (2):
  - Teva Investigational Site 761, Taipei
  - Teva Investigational Site 763, Taoyuan District
- Thailand (3):
  - Teva Investigational Site 780, Bangkok
  - Teva Investigational Site 782, Bangkok
  - Teva Investigational Site 784, Nakhon Ratchasima
- Ukraine (12):
  - Teva Investigational Site 621, Dnipropetrovsk
  - Teva Investigational Site 629, Donetsk
  - Teva Investigational Site 630, Ivano-Frankivsk
  - Teva Investigational Site 620, Kharkiv
  - Teva Investigational Site 633, Kharkiv
  - Teva Investigational Site 622, Kyiv
  - Teva Investigational Site 623, Kyiv
  - Teva Investigational Site 624, Kyiv
  - Teva Investigational Site 625, Kyiv
  - Teva Investigational Site 626, Vinnytsia
  - Teva Investigational Site 631, Zaporizhzhia
  - Teva Investigational Site 632, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1052 patients with eosinophilic asthma at 201 centers in 30 countries were enrolled in this study.
Pre-assignment Details: Four hundred-eighty (46%) patients received reslizumab for the first time in Study 3085, having previously received placebo in Studies 3081, 3082, or 3083.
Groups:
- Previous Placebo-Treated Subpopulation: The subpopulation of particpants who were treated with placebo in the previous double-blind studies. These participants were treated with resllizumab 3.0 mg/kg intravenously once every 4 weeks ( +-7 days) for up to 24 months in this study.
- Previous Reslizumab-Treated Subpopulation: The subpopulation of particpants who were treated with reslizumab at a variety of dosages in the previous double-blind studies. These participants were treated with resllizumab 3.0 mg/kg intravenously once every 4 weeks ( +-7 days) for up to 24 months in this study.
Period: Overall Study
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation
Started | 481 | 571
Safety Analysis Set | 480 (One patient was enrolled but not treated.) | 571
Completed | 15 (Completed study includes completion of the 104 week treatment phase and the 90-day follow-up.) | 35 (Completed study includes completion of the 104 week treatment phase and the 90-day follow-up.)
Not Completed | 466 | 536
Not completed — Adverse Event | 6 | 11
Not completed — Lack of Efficacy | 4 | 5
Not completed — Withdrawal by Subject | 26 | 32
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 4 | 4
Not completed — Non-compliance to study procedures | 0 | 1
Not completed — Non-compliance to study medications | 1 | 0
Not completed — Sponsor closure of study | 420 | 476
Not completed — Other | 3 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Total
Number analyzed (Participants) | 481 | 571 | 1052
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (14.53) | 47.1 (13.58) | 47.2 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 332 | 646
  Male | 167 | 239 | 406
Race/Ethnicity, Customized [Number; unit: participants]
  White | 371 | 437 | 808
  Black | 22 | 22 | 44
  Asian | 39 | 48 | 87
  American Indian or Alaskan Native | 4 | 6 | 10
  Pacific Islander | 1 | 1 | 2
  Other | 44 | 57 | 101
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 83 | 118 | 201
  Non-Hispanic or Latino | 187 | 178 | 365
  Non-Hispanic and non-Latino | 208 | 272 | 480
  Unknown | 3 | 3 | 6
Weight [Mean (Standard Deviation); unit: kg] — n=466, 555,1021
  kg | 75.4 (16.67) | 76.5 (17.85) | 76.0 (17.32)
Height [Mean (Standard Deviation); unit: cm] — n=463, 555, 1018
  cm | 165.3 (10.03) | 166.0 (9.96) | 165.7 (9.99)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — n=463, 555, 1018
  kg/m^2 | 27.6 (5.42) | 27.7 (6.04) | 27.7 (5.77)
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] | 2.096 (0.7856) | 2.285 (0.8222) | 2.199 (0.8108)
% Predicted Expiratory Volume In 1 Second [Mean (Standard Deviation); unit: percentage of predicted FEV1] | 70.739 (19.7560) | 75.116 (19.9404) | 73.115 (19.9664)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: liters] | 3.163 (1.0357) | 3.366 (1.0779) | 3.273 (1.0632)
Forced Expiratory Flow at 25% to 75% Forced Vital Capacity (FEF 25%-75%) [Mean (Standard Deviation); unit: liters/second] — n= 478, 568, 1046
  liters/second | 1.467 (0.8890) | 1.634 (0.9045) | 1.558 (0.9009)
Asthma Control Questionnaire (ACQ) [Mean (Standard Deviation); unit: units on a scale] — The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A higher score is an indication of poorer asthma control.
  n= 480, 571, 1051
  units on a scale | 1.832 (1.0912) | 1.450 (0.9870) | 1.624 (1.0527)
Asthma Quality of Life Questionnaire (AQLQ) [Mean (Standard Deviation); unit: units on a scale] — The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses.
  n= 476, 569, 1045
  units on a scale | 5.170 (1.2160) | 5.496 (1.1431) | 5.347 (1.1875)
Asthma Symptom Utility Index (ASUI) [Mean (Standard Deviation); unit: units on a scale] — The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control.
  n= 186, 191, 377
  units on a scale | 0.803 (0.1910) | 0.861 (0.1479) | 0.832 (0.1728)
Blood Eosinophil Count [Mean (Standard Deviation); unit: 10^9 blood eosinophil/L] | 0.528 (0.3792) | 0.078 (0.1480) | 0.284 (0.3577)
Used Beta Agonist in Past 3 Days [Number; unit: participants] — Usage of inhaled corticosteroids/long-acting beta-agonists and usage of oral corticosteroids.
  n= 480, 571, 1051
  participants
    Yes | 300 | 297 | 597
    No | 180 | 274 | 454
Daily average number of puffs in past 3 days [Mean (Standard Deviation); unit: puffs/day] — n= 475, 554, 1029
  puffs/day | 2.130 (2.4996) | 1.568 (2.3982) | 1.827 (2.4604)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events
Description: An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 (post-dose) to Week 65. The endpoint for adverse events was the last postbaseline observation, which included the 90 day follow-up visit.
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
participants
  At least 1 AE | 359 | 385 | 744
  Severe AE | 31 | 47 | 78
  Treatment-related AE | 49 | 41 | 90
  AE causing patient discontinuation | 6 | 12 | 18
  Serious AE | 33 | 45 | 78
  Death | 1 | 2 | 3
  AE up to follow-up period | 344 | 367 | 711
  AE during follow-up period | 78 | 82 | 160

2. Primary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Abnormal Lab Values
Description: Data represents participants with potentially clinically significant (PCS) abnormal serum chemistry, hematology, and urinalysis values on any of the during treatment lab analyses.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Creatinine: >=177 μmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * Aspartate aminotransferase: >=3*upper limit of normal (ULN). Normal range is 10-43 U/L
  * Alanine aminotransferase: >=3*ULN. Normal range is 10-40 U/L
  * GGT = gamma-glutamyl transpeptidase: >= 3*upper limit of normal. Normal range is 5-49 U/L.
  * Total bilirubin: >=34.2 μmol/L
  * White blood cells- low: <=3.0*10^9/L
  * White blood cells-high: >=20*10^9/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 L/L
  * Platelets: >=700*10^9/L
  * Absolute neutrophil count: <=1.0*10^9/L
  * Eosinophils: >=10
  * Urinalysis: ketones, blood, glucose, and total protein: >=2 unit increase from baseline
Time Frame: Weeks 4, 8, 24 and 48
Population: Safety analysis set, including participants who contributed to the analysis
Measure: Number; unit: participants
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 477 | 567 | 1044
participants
  Blood urea nitrogen | 13 | 10 | 23
  Creatinine | 3 | 2 | 5
  Uric acid | 8 | 5 | 13
  Aspartate aminotransferase | 6 | 5 | 11
  Alanine aminotransferase | 7 | 7 | 14
  GGT | 24 | 15 | 39
  Total bilirubin | 3 | 3 | 6
  White blood cells- low | 10 | 8 | 18
  White blood cells- high | 2 | 1 | 3
  Hemoglobin | 10 | 9 | 19
  Hematocrit | 13 | 13 | 26
  Platelets | 1 | 1 | 2
  Absolute neutrophil count | 7 | 7 | 14
  Eosinophils | 24 | 27 | 51
  Ketones in urine | 15 | 9 | 24
  Blood (hemaglobin) in urine | 52 | 55 | 107
  Glucose in urine | 22 | 32 | 54
  Total protein in urine | 71 | 85 | 156

3. Secondary Outcome: Forced Expiratory Volume In 1 Second (FEV1) at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma obtained from pulmonary function tests. It is the volume of air expired in the first second of a forced expiration using a spirometer.
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
liters
  Week 4 (n=457, 552, 1009) | 2.155 (0.7636) | 2.277 (0.7999) | 2.222 (0.7857)
  Week 8 (n=437, 518, 955) | 2.162 (0.7966) | 2.270 (0.8179) | 2.220 (0.8096)
  Week 12 (n=426, 499, 925) | 2.171 (0.7690) | 2.267 (0.8114) | 2.223 (0.7932)
  Week 16 (n=418, 488, 906) | 2.169 (0.7761) | 2.267 (0.8101) | 2.222 (0.7957)
  Week 24 (n=386, 458, 844) | 2.188 (0.7966) | 2.289 (0.8032) | 2.243 (0.8013)
  Week 36 (n=291, 354, 645) | 2.234 (0.8240) | 2.278 (0.8133) | 2.258 (0.8178)
  Week 48 (n=198, 250, 448) | 2.167 (0.7905) | 2.336 (0.8189) | 2.261 (0.8099)
  Week 60 (n=101, 143, 244) | 2.234 (0.9214) | 2.360 (0.8292) | 2.308 (0.8689)
  Week 72 (n=56, 105, 161) | 2.424 (0.9093) | 2.367 (0.8150) | 2.387 (0.8466)
  Week 84 (n=45, 88, 133) | 2.496 (0.8496) | 2.384 (0.8411) | 2.422 (0.8425)
  Week 96 (n=23, 46, 69) | 2.748 (0.8963) | 2.383 (0.7737) | 2.505 (0.8283)
  End of study (n=28, 54, 82) | 2.505 (0.9386) | 2.237 (0.8736) | 2.329 (0.8997)
  Endpoint (n=478, 569, 1047) | 2.174 (0.7798) | 2.273 (0.8127) | 2.228 (0.7989)

4. Secondary Outcome: Percent Predicted Forced Expiratory Volume In 1 Second (% Predicted FEV1) at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: The percent predicted FEV1 is the ratio of the volume of air expired in the first second of a forced expiration to the patient's predicted FEV based on a similar population without asthma. Percent predicted lung function values were transcribed directly from the lung function report to the CRF, without any calculation by Teva.
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
percentage of predicted FEV1
  Week 4 (n=457, 552, 1009) | 73.295 (19.7933) | 74.808 (19.1560) | 74.123 (19.4521)
  Week 8 (n=437, 518, 955) | 73.056 (19.9848) | 74.765 (20.3570) | 73.983 (20.1949)
  Week 12 (n=426, 499, 925) | 73.797 (19.2586) | 74.690 (19.8973) | 74.279 (19.6002)
  Week 16 (n=418, 488, 906) | 73.797 (19.5962) | 74.668 (20.2025) | 74.266 (19.9188)
  Week 24 (n=386, 458, 844) | 74.284 (19.5601) | 75.208 (19.9621) | 74.785 (19.7729)
  Week 36 (n=291, 354, 645) | 74.805 (20.5634) | 75.487 (20.4589) | 75.179 (20.4930)
  Week 48 (n=198, 250, 448) | 73.654 (19.9535) | 76.627 (19.8890) | 75.313 (19.9500)
  Week 60 (n=101, 143, 244) | 74.511 (22.5211) | 76.613 (20.2416) | 75.743 (21.1950)
  Week 72 (n=56, 105, 161) | 76.856 (20.1821) | 76.812 (17.1937) | 76.827 (18.2256)
  Week 84 (n=45, 88, 133) | 79.017 (18.5149) | 77.945 (18.4383) | 78.308 (18.4011)
  Week 96 (n=23, 46, 69) | 83.245 (14.9074) | 76.746 (16.2345) | 78.912 (15.9949)
  End of study (n=28, 54, 82) | 79.672 (18.6997) | 70.633 (20.2554) | 73.719 (20.0902)
  Endpoint (n=478, 569, 1047) | 74.195 (19.8134) | 75.107 (19.8530) | 74.690 (19.8307)

5. Secondary Outcome: Forced Vital Capacity (FVC) at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: The FVC is the volume of air that can be forcibly blown out after full inspiration, measured in liters.
  .
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
liters
  Week 4 (n=457, 552, 1009) | 3.222 (0.9929) | 3.372 (1.0619) | 3.304 (1.0334)
  Week 8 (n=437, 518, 955) | 3.226 (1.0228) | 3.358 (1.0836) | 3.297 (1.0577)
  Week 12 (n=426, 499, 925) | 3.238 (0.9788) | 3.339 (1.0584) | 3.292 (1.0232)
  Week 16 (n=418, 488, 906) | 3.238 (0.9949) | 3.349 (1.0835) | 3.298 (1.0444)
  Week 24 (n=386, 458, 844) | 3.233 (1.0095) | 3.369 (1.0709) | 3.307 (1.0449)
  Week 36 (n=291, 353, 644) | 3.324 (1.0571) | 3.346 (1.0416) | 3.336 (1.0479)
  Week 48 (n=198, 250, 448) | 3.229 (1.0334) | 3.414 (1.0348) | 3.332 (1.0371)
  Week 60 (n=101, 143, 244) | 3.323 (1.1874) | 3.422 (1.0428) | 3.381 (1.1037)
  Week 72 (n=56, 105, 161) | 3.500 (1.1839) | 3.398 (1.0795) | 3.434 (1.1143)
  Week 84 (n=45, 88, 133) | 3.606 (1.1403) | 3.406 (1.1535) | 3.474 (1.1487)
  Week 96 (n=23, 46, 69) | 3.849 (1.2342) | 3.381 (1.1145) | 3.537 (1.1680)
  End of study (n=28, 54, 82) | 3.524 (1.1842) | 3.321 (1.2443) | 3.390 (1.2206)
  Endpoint (n=478, 569, 1047) | 3.250 (1.0194) | 3.355 (1.0675) | 3.307 (1.0466)

6. Secondary Outcome: Forced Expiratory Flow at 25% to 75% Forced Vital Capacity (FEF 25%-75%) at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: The FEF 25%-75% is the force expiratory flow at 25% to 75% of the Forced Vital Capacity (FVC), measured in liters/second
  .
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
liters/second
  Week 4 (n=446, 545, 991) | 1.558 (0.9363) | 1.614 (0.9055) | 1.589 (0.9195)
  Week 8 (n=429, 513, 942) | 1.546 (0.9279) | 1.618 (0.9255) | 1.585 (0.9268)
  Week 12 (n=418, 494, 912) | 1.587 (0.9833) | 1.624 (0.9367) | 1.607 (0.9580)
  Week 16 (n=408, 483, 891) | 1.561 (0.9427) | 1.620 (0.9068) | 1.593 (0.9234)
  Week 24 (n=377, 453, 830) | 1.619 (0.9967) | 1.637 (0.9227) | 1.629 (0.9565)
  Week 36 (n=285, 349, 634) | 1.642 (1.1087) | 1.650 (0.9193) | 1.646 (1.0080)
  Week 48 (n=191, 249, 440) | 1.628 (1.0408) | 1.691 (0.9450) | 1.664 (0.9871)
  Week 60 (n=99, 143, 242) | 1.605 (1.0869) | 1.791 (1.1508) | 1.715 (1.1265)
  Week 72 (n=56, 105, 161) | 1.810 (1.0239) | 1.766 (1.0341) | 1.781 (1.0276)
  Week 84 (n=45, 88, 133) | 1.848 (0.9047) | 1.892 (1.1499) | 1.877 (1.0700)
  Week 96 (n=23, 46, 69) | 2.120 (1.0597) | 1.942 (1.0453) | 2.001 (1.0457)
  End of study (n=28, 54, 82) | 1.939 (1.1105) | 1.639 (0.9079) | 1.741 (0.9854)
  Endpoint (n=468, 563, 1031) | 1.546 (0.9041) | 1.629 (0.9300) | 1.592 (0.9188)

7. Secondary Outcome: Average Daily Use of Short-Acting Beta-Agonist (SABA)Therapy at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: SABA are used for quick relief of asthma symptoms. To measure SABA use, at each clinical visit participants were asked to recall their usage of SABA therapy within the last 3 days of the scheduled visit. If usage was confirmed, the number of puffs used was recorded. For the purpose of summaries, an average daily usage was evaluated by dividing the total number of puffs recorded over 3 days by 3.
  .
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: # puffs/day
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
# puffs/day
  Week 4 (n=276, 323, 599) | 2.5 (2.42) | 2.4 (2.45) | 2.5 (2.43)
  Week 8 (n=258, 302, 560) | 2.4 (2.28) | 2.4 (2.62) | 2.4 (2.46)
  Week 12 (n=251, 278, 529) | 2.6 (2.07) | 2.4 (2.50) | 2.5 (2.30)
  Week 16 (n=244, 261, 505) | 2.5 (2.30) | 2.2 (2.29) | 2.4 (2.30)
  Week 24 (n=211, 243, 454) | 2.6 (2.55) | 2.3 (2.46) | 2.4 (2.51)
  Week 36 (n=160, 174, 334) | 2.4 (2.27) | 2.3 (2.64) | 2.3 (2.47)
  Week 48 (n=111, 121, 232) | 2.2 (2.28) | 2.4 (2.54) | 2.3 (2.42)
  Week 60 (n=50, 64, 114) | 2.1 (2.19) | 2.5 (3.30) | 2.3 (2.86)
  Week 72 (n=29, 47, 76) | 2.1 (2.19) | 1.8 (1.88) | 1.9 (1.99)
  Week 84 (n=19, 35, 54) | 2.0 (1.57) | 2.4 (2.38) | 2.2 (2.12)
  Week 96 (n=14, 26, 40) | 1.8 (1.41) | 1.7 (1.57) | 1.8 (1.50)
  End of study (n=16, 23, 39) | 2.1 (1.76) | 2.7 (1.99) | 2.4 (1.90)
  Endpoint (n=390, 453, 843) | 2.2 (2.20) | 2.2 (4.09) | 2.2 (3.35)

8. Primary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Vital Signs Values
Description: Data represents participants with PCS vital sign values during any of the during treatment visits or the follow-up visit.
  Significance criteria
  * Sitting heart rate-high: >100 and increase of >= 30 beats/min (all ages)
  * Sitting heart rate-low: <50 and decrease of >=30 beats/min
  * Sitting systolic blood pressure (BP)-high: >130 and increase of >=30 mmHg (ages 12-17)
  * Systolic BP-low: <90 and decrease of >=30 mmHg (ages >=18)
  * Systolic BP-high: >160 and increase of >=30 mmHg (ages >=18)
  * Sitting diastolic BP-low: <55 and decrease of >=12 mmHg (ages 12-17)
  * Diastolic BP-high: >85 and increase of >=12 mmHg (ages 12-17)
  * Diastolic BP-low: <50 and decrease of >=12 mmHg (ages >=18)
  * Diastolic BP-high: >100 and increase of >=12 mmHg (ages >=18)
  * Respiration rate: >20 and increase of >=10 breaths/minute (ages 12-17)
  * Respiration rate: >24 and increase of >=10 breaths/minute (ages >=18)
  * Body temperature-low: <96.5° Fahrenheit (all ages)
  * Body temp-high: >100.5° F (all ages)
Time Frame: Week 4 to Week 65
Population: Safety analysis set, including participants who contributed to the analysis
Measure: Number; unit: participants
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 478 | 569 | 1047
participants
  Heart rate - high (ages 12-17) | 1 | 2 | 3
  Heart rate - low (ages >=18) | 2 | 1 | 3
  Heart rate - high (ages >=18) | 8 | 8 | 16
  Systolic BP - high (ages 12-17) | 0 | 1 | 1
  Systolic BP - low (ages >=18) | 1 | 0 | 1
  Systolic BP - high (ages >=18) | 8 | 8 | 16
  Diastolic BP - low (ages 12-17) | 1 | 1 | 2
  Diastolic BP - high (ages 12-17) | 2 | 1 | 3
  Diastolic BP - low (ages >=18) | 2 | 4 | 6
  Diastolic - high (ages >=18) | 13 | 12 | 25
  Respiration rate - high (ages 12-17) | 0 | 1 | 1
  Respiration rate - high (ages >=18) | 6 | 2 | 8
  Body temperature - low (ages 12-17) | 3 | 3 | 6
  Body temperature - high (ages 12-17) | 0 | 1 | 1
  Body temperature - low (ages >=18) | 102 | 121 | 223
  Body temperature - high (ages >=18) | 3 | 1 | 4

9. Secondary Outcome: Asthma Symptom Utility Index (ASUI) Score at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control.
  .
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
units on a scale
  Week 4 (n=456, 552, 1008) | 0.831 (0.1829) | 0.844 (0.1631) | 0.838 (0.1724)
  Week 8 (n=436, 514, 950) | 0.843 (0.1663) | 0.851 (0.1596) | 0.847 (0.1626)
  Week 12 (n=426, 500, 926) | 0.839 (0.1752) | 0.854 (0.1578) | 0.847 (0.1661)
  Week 16 (n=416, 486, 902) | 0.845 (0.1690) | 0.856 (0.1659) | 0.851 (0.1673)
  Week 24 (n=386, 458, 844) | 0.844 (0.1720) | 0.859 (0.1602) | 0.852 (0.1658)
  Week 36 (n=291, 354, 645) | 0.844 (0.1821) | 0.867 (0.1536) | 0.857 (0.1673)
  Week 48 (n=198, 251, 449) | 0.851 (0.1699) | 0.856 (0.1705) | 0.854 (0.1701)
  Week 60 (n=100, 146, 246) | 0.869 (0.1573) | 0.865 (0.1513) | 0.866 (0.1534)
  Week 72 (n=56, 105, 161) | 0.876 (0.1346) | 0.858 (0.1509) | 0.865 (0.1453)
  Week 84 (n=45, 87, 132) | 0.884 (0.1460) | 0.868 (0.1541) | 0.873 (0.1510)
  Week 96 (n=23, 46, 69) | 0.822 (0.2036) | 0.836 (0.1729) | 0.832 (0.1823)
  End of study (n=28, 55, 83) | 0.877 (0.0979) | 0.840 (0.2053) | 0.853 (0.1767)
  Endpoint (n=478, 569, 1047) | 0.843 (0.1679) | 0.850 (0.1661) | 0.847 (0.1669)

10. Secondary Outcome: Asthma Control Questionnaire (ACQ) at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, End of Study and Endpoint
Description: The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A higher score is an indication of poorer asthma control.
Time Frame: Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, 96, end of study and endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
units on a scale
  Week 4 (n=456, 552, 1008) | 1.546 (1.0154) | 1.429 (0.9573) | 1.482 (0.9852)
  Week 8 (n=437, 517, 954) | 1.446 (0.9805) | 1.392 (0.9729) | 1.417 (0.9762)
  Week 12 (n=426, 500, 926) | 1.459 (1.0004) | 1.360 (0.9320) | 1.405 (0.9648)
  Week 16 (n=416, 487, 903) | 1.444 (1.0016) | 1.305 (0.9299) | 1.369 (0.9655)
  Week 24 (n=386, 458, 844) | 1.436 (1.0135) | 1.299 (0.9497) | 1.362 (0.9812)
  Week 36 (n=291, 353, 644) | 1.425 (1.0189) | 1.282 (0.9331) | 1.347 (0.9746)
  Week 48 (n=198, 250, 448) | 1.408 (0.9699) | 1.297 (0.9810) | 1.346 (0.9766)
  Week 60 (n=100, 143, 243) | 1.284 (0.9739) | 1.297 (0.9432) | 1.292 (0.9540)
  Week 72 (n=56, 105, 161) | 1.283 (0.9176) | 1.231 (0.8295) | 1.249 (0.8587)
  Week 84 (n=45, 87, 132) | 1.143 (0.9020) | 1.209 (0.9186) | 1.186 (0.9100)
  Week 96 (n=23, 46, 69) | 1.323 (0.9862) | 1.391 (0.9559) | 1.369 (0.9594)
  End of study (n=28, 54, 82) | 1.061 (0.7653) | 1.437 (0.9750) | 1.308 (0.9216)
  Endpoint (n=478, 569, 1047) | 1.450 (0.9901) | 1.389 (0.9637) | 1.417 (0.9759)

11. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) Total Score at Weeks 24, 48, 72, 96, End of Study and Endpoint
Description: The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses. Five of the activity questions were "patient-specific," which means that each patient identified and scored 5 activities in which the patient was limited by asthma; these 5 activities were identified at the first visit and retained for all subsequent follow-up visits.
Time Frame: Weeks 24, 48, 72, 96, End of Study and Endpoint
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 480 | 571 | 1051
units on a scale
  Week 24 (n=382, 452, 834) | 5.551 (1.1558) | 5.691 (1.0651) | 5.627 (1.1091)
  Week 48 (n=193, 249, 442) | 5.602 (1.1180) | 5.725 (1.0818) | 5.672 (1.0982)
  Week 72 (n=56, 106, 162) | 5.808 (1.0002) | 5.809 (1.0235) | 5.809 (1.0124)
  Week 96 (n=23, 46, 69) | 5.585 (1.1422) | 5.809 (1.1340) | 5.734 (1.1333)
  End of study (n=28, 55, 83) | 5.956 (0.9431) | 5.765 (1.2361) | 5.829 (1.1434)
  Endpoint (n=472, 558, 1030) | 5.535 (1.1690) | 5.631 (1.1334) | 5.587 (1.1503)

12. Secondary Outcome: Participants With a Positive Anti-Reslizumab Antibody Status at Baseline, Weeks 24, 48, 72, 96, End of Study, Endpoint and Overall
Description: Blood samples were collected for the determination of anti-drug antibody (ADAs) before study drug infusion at baseline and every 24 weeks until end of treatment visit or early withdrawal. Serum samples were analyzed by Teva (Teva Biopharmaceuticals USA, Rockville, Maryland, USA) using a validated homogeneous solution based bridging enzyme linked immune sorbent assay (Mikulsis et al 2011, Qui et al 2010). The analysis of anti-reslizumab antibody in patient serum consists of 3 tiers of assays for screening, confirmation, and titer analysis. If a participant had a treatment-emergent ADA response (ie, ADA positive at any of the postdose time points but negative at the predose time point) or if there was a treatment-boosted ADA response (defined as a greater than 4-fold increase from a positive baseline ADA response (Shankar et at 2014), the participant was classified as overall ADA positive.
  Predose samples for the reslizumab-experienced participants came from the previous studies.
Time Frame: Baseline, Weeks 24, 48, 72, 96, End of Study, Endpoint and Overall
Population: Safety analysis set of participants with assessments at stated timeframes
Measure: Number; unit: participants
Arm/Group | Previous Placebo-Treated Subpopulation | Previous Reslizumab-Treated Subpopulation
Number analyzed (Participants) | 480 | 571
participants
  Overall (n=466, 548) | 24 | 25
  Baseline (n=442, 541) | 16 | 24
  Week 24 (n=382, 445) | 12 | 13
  Week 48 (n=187, 247) | 9 | 7
  Week 72 (n=56, 104) | 4 | 4
  Week 96 (n=24, 48) | 3 | 1
  End of study (n=142, 52) | 4 | 1
  Endpoint (n=466, 545) | 12 | 17

ADVERSE EVENTS:
Time Frame: Day 1 (post-dose) to Week 65. The endpoint for adverse events was the last postbaseline observation, which included the 90 day follow-up visit.
Arm/Group | Reslizumab 3.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 78/1051
Other Adverse Events (participants affected / at risk) | 519/1051
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 3.0 mg/kg (N=1051)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Suprapubic pain (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis pneumococcal (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (4)
Suicide attempt (Psychiatric disorders) | 2 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 (24)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 3.0 mg/kg (N=1051)
Bronchitis (Infections and infestations) | 62 (77)
Nasopharyngitis (Infections and infestations) | 150 (226)
Sinusitis (Infections and infestations) | 77 (114)
Upper respiratory tract infection (Infections and infestations) | 107 (141)
Headache (Nervous system disorders) | 73 (106)
Asthma (Respiratory, thoracic and mediastinal disorders) | 301 (563)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.